CLINICAL TRIAL: NCT05197127
Title: Implementing a Robotic Hip Assist-based Mobility Intervention for Older Adults With Frailty
Brief Title: Efficacy of Samsung GEMS-H Device Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director, Max Nader Lab, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hip Exoskeleton Older Adult
Record Dates: First submitted 2021-12-17; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Geriatrics
Keywords: Geriatrics; Gait Training; Exoskeleton; Fall Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Walking Group (Experimental): Twelve participants over 65 years old completed a total of twelve 30-minute gait training sessions over a period of 4-6 weeks using the GEMS-H. All gait training sessions were completed in the community spaces at a senior living community. Gait training included dynamic over-ground walking (both self-selected and fast-paced),variable conditions of multi-directional walking, and training on ramps, stairs, and obstacle negotiation.
  Interventions: Device: exoskeleton-based gait training

INTERVENTIONS:
Device: exoskeleton-based gait training — Gait training included dynamic over-ground walking (both self-selected and fast-paced), variable conditions of multi-directional walking, and training on ramps, stairs, and obstacle negotiation.

SUMMARY:
The purpose of this study is to evaluate the feasibility of using Samsung robotic hip assist-based mobility intervention for older adults with frailty.

The specific aims of this project are:

Aim 1 Will investigate the feasibility of the Samsung robotic hip assist-based mobility intervention on gait function, sedentary time, and fall risk.

Hypothesis: A 6-week robotic device-based mobility intervention will improve locomotor gait function, sedentary time, and fall risk.

DETAILED DESCRIPTION:
Twelve individuals above the age of 65 years old were recruited to participate in twelve sessions that occurred 2-3 times per week over a 4-6 week period using the GEMS-H. In addition to selecting individuals over the age of 65, qualifying participants also had to be able to walk with or without an assistive device for greater than ten feet. Medical clearance was obtained from each participant's primary physician prior to training with the device.

Gait training included dynamic over-ground walking (both self-selected and fast-paced), variable conditions of multidirectional walking, and training on ramps, stairs, and obstacle negotiation. All training was done under the supervision of a trained physical therapist. The amount of assistance and resistance torque provided by the hip motors of the GEMS-H was personalized according to each participant's specific abilities and self-reported tolerance/comfort throughout each session. These modifications followed a training progression model of increasing resistance and decreasing assistance over the course of the twelve sessions to maximize the challenge and improve strength and endurance in each participant.

ELIGIBILITY:
Inclusion Criteria:

* They are primarily English speaking
* > 65 years of age
* Able to walk with or without an assistive device >10 feet
* Able to obtain medical clearance from the participant's primary physician
* We will not include any special populations in this study

Exclusion Criteria:

* Cannot comprehend or provide inform consent
* Unable to fit the device within the hip frame size of310mm-380mm (approximately 12-15 inches)
* Other weight and length limitations that restrict the proper fit of the device
* Any significant neurological diagnosis impacting safe use of the device

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test Speed | 0 weeks and through study completion (average of 4-6 weeks)
  Average walking speed measured over 10 meters, tested at self selected velocity and fast velocity
Change in 6 minute walk test distance | 0 weeks and through study completion (average of 4-6 weeks)
  distance in meters covered in six minutes
Change in Berg Balance Scale Score | 0 weeks and through study completion (average of 4-6 weeks)
  Total score across 14 items in the Berg Balance Scale, scored 0-56 (maximum score is 56)
Change in Functional Gait Assessment Score | 0 weeks and through study completion (average of 4-6 weeks)
  Total score across 10 items in the Functional Gait Assessment, scored 0-30 (maximum score is 30)
Change in 5 Times Sit-to-Stand Time | 0 weeks and through study completion (average of 4-6 weeks)
  The time required to stand up and sit down from a chair five times without assistance

SECONDARY OUTCOMES:
Change in Sedentary Bouts per day | 0 weeks and through study completion (average of 4-6 weeks)
  Using a wearable sensor, we measured the number of sedentary bouts greater than 3 minutes per day

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PHD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jayaraman C, Embry KR, Mummidisetty CK, Moon Y, Giffhorn M, Prokup S, Lim B, Lee J, Lee Y, Lee M, Jayaraman A. Modular hip exoskeleton improves walking function and reduces sedentary time in community-dwelling older adults. J Neuroeng Rehabil. 2022 Dec 30;19(1):144. doi: 10.1186/s12984-022-01121-4. PMID 36585676